CLINICAL TRIAL: NCT00926614
Title: 48 Week Pilot Trial Assessing the Efficacy of Pioglitazone, Atorvastatin, Pegasys and Weight Based Ribavirin in Chronic Hepatitis C, Genotype 1 Patients Who Have Previously Relapsed or Did Not Respond to PegInterferon /Ribavirin Therapy
Brief Title: Efficacy of Actos Lipitor Pegasys & Ribavirin in CHC GT 1 Patients Who Relapsed or Nonresponded to Peg/Riba
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephen A Harrison, Principal Investigator, Brooke Army Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.2008.153
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hepatitis c
Keywords: GT1; HCV; non responder; relapser
MeSH Terms: conditions — Hepatitis C | interventions — Pioglitazone; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pioglitizone and Atorvastatin (Experimental): Pioglitazone and Atorvastatin added to standard of care Pegasys and weight based ribavirin
  Interventions: Drug: pioglitazone (Actos); Drug: atorvastatin (Lipitor)

INTERVENTIONS:
Drug: pioglitazone (Actos) — pioglitazone 30 mg qd for 30 days, then increase to 45 mg
  Other Names: Actos
Drug: atorvastatin (Lipitor) — atorvastatin 40 mg for 30 days then increase to 80 mg daily
  Other Names: Lipitor

SUMMARY:
The aim of the study will be to determine if an insulin sensitizing thiazolidinedione plus a lipid lowering agent (statin) improves sustained virologic response rates in patients who have previously not responded or relapsed on standard pegylated interferon and ribavirin therapy.

DETAILED DESCRIPTION:
The study will evaluate the use of atorvastatin and pioglitazone in the pre-treatment of insulin resistance and lipid levels prior to the addition of pegylated interferon and ribavirin for chronic hepatitis C (CHC). If improvement is seen in insulin resistance patients may then be in a position to respond more favorably to current antiviral therapy consisting of pegylated interferon and ribavirin.

This study could demonstrate the value of pretreating and continuing treatment for insulin resistance with pioglitazone in CHC, genotype 1 patients who have previously not responded or relapsed to prior pegylated interferon and ribavirin treatment. Changes in lipids are not a primary or secondary endpoint in this study.

ELIGIBILITY:
Inclusion Criteria:

* GT 1 previously treated with pegylated interferon & ribavirin & either non-responded or relapsed after cessation of therapy
* Insulin resistance
* Compensated liver disease

  * WBC < 3,000/ mm3
  * Neutrophil count < 1,500/mm3
  * Platelets < 65,000/ mm3
  * Albumin > 3 gm/dL

Exclusion Criteria:

* Participants on metformin or other thiazolidinedione must have 3month wash-out period
* Women who are pregnant or breast-feeding
* Males with pregnant partners
* Co-infection with HAV, HBV, or HIV
* Ophthalmic abnormalities such as severe retinopathy
* Poorly controlled thyroid dysfunction
* Serum creatinine concentration > 1.5 times ULN
* Severe psychiatric or neuropsychiatric disorders
* History of alcoholism or drug addiction 1 year prior to screening
* Seizure disorders not controlled with medication
* Significant cardiovascular dysfunction within the past 12 months
* Chronic pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement is seen in insulin resistance patients to be in a position to respond more favorably to current antiviral therapy consisting of pegylated interferon and ribavirin. | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Harrison, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States